CLINICAL TRIAL: NCT00117897
Title: An Open-Label, Randomized, Parallel, Phase II Study of CHOP Chemotherapy and Rituximab Administered Every 14 Days, With Pegfilgrastim or Filgrastim Support, for the Treatment of Subjects With Non-Hodgkin's Lymphoma
Brief Title: Treatment for Subjects With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010157
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: non-Hodgkin's lymphoma; R-CHOP-14; pegfilgrastim; neutropenia, clinical trial; haematopoietic growth factor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neutropenia | interventions — pegfilgrastim; Filgrastim

INTERVENTIONS:
Drug: pegfilgrastim
Drug: Filgrastim

SUMMARY:
This multicenter, open-label, randomized, parallel study was designed to evaluate whether a single fixed-dose subcutaneous (SC) administration of pegfilgrastim or daily administration of Filgrastim for absolute neutrophil count (ANC) support would assist in allowing the planned dose-on-time (PDOT) of cyclophosphamide, doxorubicin, vincristine, prednisolone (CHOP) chemotherapy with Rituximab every 14 days in subjects with aggressive B-cell Non-Hodgkin's Lymphoma by reducing the duration of neutropenia and incidence of febrile neutropenia.

ELIGIBILITY:
Inclusion Criteria: - Histologically proven aggressive B-cell Non-Hodgkin's lymphoma (IWF classification D-H) with: - Bone marrow involvement less than 30% demonstrated by aspiration - Age-adjusted International Prognostic Index (IPI) 0-2 - Measurable or evaluable disease - ECOG performance status 0-2 - Life expectancy greater than or equal to 12 weeks - Absolute neutrophil count greater than 1.5 x 109/L - Platelet count greater than 100 x 109/L - Adequate organ function (serum creatinine less than or equal to 2.0 mg/dL, SGOT/AST and SGPT/ALT less than 3 x the upper limit of normal, hemoglobin greater than or equal to 10g/dL and total serum bilirubin less than or equal to 1.5 mg/dL) - Left Ventricular Ejection Fraction (LVEF) greater than or equal to 50% at rest by MUGA or echocardiogram - Previously untreated with chemotherapy or radiotherapy - Before any study specific procedure or before study medication was administered, the subject was to give written informed consent for participation in the study Exclusion Criteria: - Burkitt's or B-lymphoblastic lymphoma - CNS involvement - Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, antiviral) within 72 hours of chemotherapy - Use of anti-hypertensives within 12 hours of start of chemotherapy - Known HIV infection - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukaemia) - Prior malignancy within the last 5 years, with the exception of surgically cured basal cell carcinoma, squamous skin cell carcinoma, or in situ carcinoma of the cervix - Prior bone marrow or stem cell transplantation - History of impaired cardiac status, e.g. severe heart disease,cardiomyopathy, or congestive heart failure - Major surgery within 2 weeks prior to randomization - Subject is evidently pregnant (e.g., positive HCG test unless termination is proven) or is breast feeding - Subject is not using adequate contraceptive precautions - Known hypersensitivity to E coli-derived products (e.g., Filgrastim,HUMULIN® Insulin, L-Asparaginase, HUMATROPE® Growth Hormone, INTRON A®) - Any psychiatric, addictive or other kind of disorder which compromised the ability of the subject to give written informed consent and/or to comply with study protocol procedures - Prior exposure to pegfilgrastim - Subject is currently enrolled in, or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving other investigational agent(s) - Subject has previously entered this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2004-02

PRIMARY OUTCOMES:
The primary objective was to provide preliminary information on the ability of pegfilgrastim or Filgrastim to support planned dose on time (PDOT) application of CHOP chemotherapy with Rituximab given every 14 days, to subjects with NHL.

SECONDARY OUTCOMES:
The proportion of chemotherapy cycles given at the PDOT in both arms.
Response rates (complete response and partial response) in both arms
The safety profile in cycles 1-6
Subject self-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20010157.pdf